CLINICAL TRIAL: NCT01966328
Title: A Safety and Efficacy Assessment of Resolvine for Treatment of Vitreomacular Attachment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeffrey S Heier (Other)
Collaborators: Kato Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jeffrey S Heier, Sponsor-Investigator, Ophthalmic Consultants of Boston
Organization: Ophthalmic Consultants of Boston (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VMA-001
Record Dates: First submitted 2013-10-14; First posted 2013-10-21 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Vitreomacular Attachment; Vitreomacular Traction; Vitreomacular Adhesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 36% Resolvine (Experimental): Patients in this arm will be given one dose of 36% Resolvine intravitreal injection, with the possibility of a second dose at Day 30
  Interventions: Drug: 36% Resolvine Intravitreal Injection
- 9% Resolvine (Active Comparator): Patients in this arm will be given one dose of 9% Resolvine intravitreal injection, with the possibility of a second dose at Day 30
  Interventions: Drug: 9% Resolvine Intravitreal Injection

INTERVENTIONS:
Drug: 36% Resolvine Intravitreal Injection — 36% Resolvine Intravitreal Injection
  Arms: 36% Resolvine
Drug: 9% Resolvine Intravitreal Injection — 9% Resolvine Intravitreal Injection
  Arms: 9% Resolvine

SUMMARY:
This research is studying the effect that Resolvine injection will have on patients with vitreomacular adhesion.

DETAILED DESCRIPTION:
This research is studying the effect that Resolvine injection will have on patients with vitreomacular adhesion. The investigators propose that intravitreal injection of Resolvine® 36% will: 1)Result in release of the vitreous adhesion to the macula in subjects with symptomatic vitreomacular attachment (VMA). 2)The Release of the VMA will create a measurable and favorable retinal change. 3) The release of vitreomacular traction may also result in visual acuity improvement within the short time frame of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18 years of age or older
2. Willing and able to return for all study visits
3. Willing and able to provide written informed consent
4. Have symptomatic VMA.
5. If both eyes are found to have Anatomic VMA the eye with lower visual acuity will be declared the study eye.

Exclusion Criteria:

1. Subjects with high myopia in the study eye (axial length greater than or equal to 26.0 millimeters by ultrasound or spherical equivalent at the spectacle plane greater than -8.0 diopters)
2. Subjects who have monocular vision or contralateral vision of 20/400 or worse BCVA in the non-study eye
3. Subjects with a history of retinal detachment or tear in the study eye
4. Subjects who have PVD in the study eye at Baseline (Grade III or greater PVD by B-scan)
5. Subjects with unstable IOP (i.e. > 30 mmHg in the past six months) or IOP of > 21 mm Hg at enrollment, under medical control. Subjects may be on topical medications to control their IOP but may not stop or start a prostaglandin type or epinephrine based drug during the study.
6. Subjects with an aphakic study eye or if pseudophakic, cataract extraction surgery less than 6 months prior to study enrollment
7. Subjects with a history of ocular trauma of any type in the study eye
8. Subjects with media opacities or abnormalities that would preclude observation of the retina in the study eye per the investigator's judgment
9. Subjects that have undergone any previous vitrectomy (either anterior or pars plana vitrectomy) in the study eye
10. Subjects with a history of cataract surgery complications in the study eye
11. Subjects that have undergone previous photocoagulation of the retina in the study eye
12. Subjects with any evidence or history of either nonproliferative or proliferative diabetic retinopathy (NPDR) or (PDR) in the study eye
13. Subjects with an anticipated need for cataract extraction in the study eye within the next 6 months
14. Subjects with congenital eye malformations
15. Subjects with recurrent uveitis or history of uveitis in either eye
16. Subjects with ongoing ocular infection or inflammation in the study eye
17. Subjects who are pregnant or nursing. Subjects of child bearing ages will undergo pregnancy testing.
18. Subjects that are currently participating in any other investigational research study
19. Subjects who are too ill to be likely to complete the entire study
20. Subjects who have undergone major surgery within the last 6 months (systemic or ocular) or who are likely to require major surgery in the upcoming 6 months
21. Subjects who are uncontrolled diabetics (HbA1/C > 10%) with significant morphological pathology at the time of enrollment
22. Subjects with macular holes Stage 2 or greater as determined by OCT, B-scan ultrasound and clinical examination
23. Subjects with epiretinal membrane (ERM) at the area of attachment as determined by OCT
24. Subjects that have received other intravitreal injection therapy within thirty (30) days of treatment with Resolvine®
25. Subjects that have received more than one Jetrea injection in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Safety of 36% Resolvine Injection versus 9% Resolvine Injection | After all patients have completed the 6 month follow-up.
  The primary objective of this study is to evaluate the safety of an active arm treated with Resolvine® 36%, which may contain up to two 100-microliter intravitreal injections, in comparison to a control arm treated with Resolvine 9%, which may contain up to two 100-microliter injections, in subjects with VMA. Cumulative adverse event rates for each arm will be evaluated.
Efficacy of 36% Resolvine Injection versus 9% Resolvine Injection | After all patients have completed the 6 month follow-up
  The primary objective of this study is to evaluate the efficacy of an active arm treated with Resolvine® 36%, which may contain up to two 100-microliter intravitreal injections, in comparison to a control arm treated with Resolvine 9%, which may contain up to two 100-microliter injections, in subjects with VMA. Efficacy will be measured by the percent of patients whose VMA has released after treatment.

SECONDARY OUTCOMES:
Inducement of PVD | After all patients have completed the 6 month follow-up
  These analyses will compare the efficacy an active arm treated with Resolvine® 36%, which may contain up to two 100-microliter intravitreal injections, to a control arm treated with Resolvine 9%, which may contain up to two 100-microliter injections, to assess inducement of a more extensive PVD over the study period as demonstrated by Trese Grade III or higher B-Scan Ultrasound and OCT.
Improved Eye Function | After all patients have completed the 6 month follow-up.
  These analyses will assess a parameter of improved eye function as calculated by either the reduction in the retinal thickness of at least 10% over baseline at Day 0 as quantified by OCT, or an improvement in visual acuity of more than 10% over baseline at day 0 as quantified by ETDRS.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Heier, MD, Principal Investigator — Ophthalmic Consultants of Boston
Locations (2):
- United States (2):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Ophthalmic Consultants of Boston, Boston, Massachusetts